CLINICAL TRIAL: NCT02836496
Title: Study 200622: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of Mepolizumab in the Treatment of Adolescent and Adult Subjects With Severe Hypereosinophilic Syndrome
Brief Title: Efficacy and Safety Study of Mepolizumab in Subjects With Severe Hypereosinophilic Syndrome (HES)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200622
Expanded Access: NCT00244686 (No longer available)
Record Dates: First submitted 2016-07-14; First posted 2016-07-19 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Hypereosinophilic Syndrome
Keywords: Safety; Mepolizumab; Hypereosinophilic syndrome; HES flare; Efficacy
MeSH Terms: conditions — Hypereosinophilic Syndrome | interventions — mepolizumab; Prednisolone; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mepolizumab (Experimental): Enrolled subjects will receive either mepolizumab 300 mg or placebo subcutaneous (SC) every 4 weeks while continuing their HES therapy.
  Interventions: Drug: Mepolizumab 300 mg; Drug: Active OCS capsules (5 mg prednisolone or prednisone); Drug: Placebo matching OCS capsules
- Placebo (Placebo Comparator): Enrolled subjects will receive either mepolizumab 300 mg or placebo SC every 4 weeks while continuing their HES therapy.
  Interventions: Drug: Placebo matching mepolizumab; Drug: Active OCS capsules (5 mg prednisolone or prednisone); Drug: Placebo matching OCS capsules

INTERVENTIONS:
Drug: Mepolizumab 300 mg — Mepolizumab is available as lyophilized powder for injection reconstituted with Sterile Water for Injection, just prior to use.
  Arms: Mepolizumab
Drug: Placebo matching mepolizumab — Placebo is available as 0.9% sodium chloride solution
  Arms: Placebo
Drug: Active OCS capsules (5 mg prednisolone or prednisone) — All subjects will be provided with 2 bottles of blinded OCS capsules, one containing 5mg OCS capsules (active OCS treatment) and a second one containing matching placebo capsules (placebo OCS treatment). These will be dispensed to each subject at each scheduled clinic visit and as needed. Subjects with an increase in blood eosinophils above the pre-specified threshold will be instructed to start blinded OCS treatment from one of the bottles provided (active treatment) unless the subject's HES therapy has already been increased due to a symptom flare within the past 2 weeks.
Drug: Placebo matching OCS capsules — All subjects will be provided with 2 bottles of blinded OCS capsules, one containing 5mg OCS capsules (active OCS treatment) and a second one containing matching placebo capsules (placebo OCS treatment). These will be dispensed to each subject at each scheduled clinic visit and as needed.A subject who does not reach the pre-specified blood eosinophil threshold with a similar blood draw date will be selected to initiate a placebo OCS treatment in a blinded manner, unless the subject's HES therapy has already been increased due to a symptom flare within the past 2 weeks.

SUMMARY:
Mepolizumab is a humanized monoclonal antibody. In conditions where eosinophilia is considered to play an important part in the pathology, including eosinophilic asthma, HES, and eosinophilic granulomatosis with polyangiitis, a consistent reduction in blood eosinophil counts is observed in association with mepolizumab administration, with concomitant clinical improvement. This is a 32-week treatment period, randomized, double-blind, placebo-controlled, parallel group, multicentre study of mepolizumab in adolescent and adult subjects with severe HES receiving standard of care (SoC) therapy. This study will demonstrate the efficacy of mepolizumab compared with placebo based on maintenance of control of HES symptoms during the treatment period. The study will comprise of a screening period of up to approximately 4 weeks followed by a 32-Week study treatment period (subjects will be randomized 1:1 to placebo or mepolizumab) and up to 8-week additional follow-up period (12 weeks after the last dose of study treatment).

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent/assent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol
* Twelve years of age or older, at the time of signing the informed consent/assent
* Subjects who have been diagnosed with HES for at least 6 months at randomization
* A history of two or more HES flares within the past 12 months prior to screening. Historical HES flares are defined as documented HES-related worsening of clinical symptoms or blood eosinophil counts requiring an escalation in therapy. At least one HES flare within the past 12 months must not be related to a decrease in HES therapy during the 4 weeks prior to the flare.
* Subjects must have blood eosinophil count >=1000 cells/µL present in the sample collected during screening (within 4 weeks prior to randomization).
* Subjects must be on a stable dose of HES therapy for the 4 weeks prior to randomization. HES therapy includes but is not limited to oral corticosteroid, immunosuppressive, and cytotoxic therapy.
* Male or female. A female subject is eligible to participate if she is not pregnant, not lactating, and either non-reproductive potential or reproductive potential and agree to use a highly effective method to avoid pregnancy from 30 days prior to the first dose of study medication and until 4 months after the last dose of study treatment.

Exclusion Criteria:

* Life-threatening HES or life-threatening HES co-morbidities: Imminently life-threatening HES disease severity such that the likelihood of death is high unless the course of the disease is interrupted within 12 weeks prior to randomization.
* Subjects who have known, pre-existing, clinically significant endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, hematological, respiratory or any other system abnormalities that are not associated with HES and are uncontrolled with standard treatment.
* Eosinophilia of unknown clinical significance
* Twelve-lead electrocardiogram (ECG) finding: QT interval corrected for heart rate (QTc) > 450 msec or QTc > 480 msec in subjects with bundle branch block or an abnormal ECG finding from the 12-lead ECG conducted at Visit 1 if considered to be clinically significant and would impact the subject's participation during the study based on the evaluation of the Investigator.
* Subjects with documented history of any clinically significant cardiac damage prior to screening that, in the opinion of the investigator, would impact the subject's participation during the study.
* Liver abnormality/disease - Alanine transaminase (ALT) >2.5x upper limit of normal (ULN) or ALT>5xULN if documented HES with liver manifestations, or bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent), or current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment). Stable chronic liver disease should generally be defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice, or cirrhosis.

NOTE: Chronic stable hepatitis B and C (e.g., presence of hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment) are acceptable if subject otherwise meets entry criteria.

* Clinical diagnosis of eosinophilic granulomatosis with polyangiitis (EGPA)
* Subjects with a history of or current lymphoma, or subjects with current malignancy or previous history of cancer in remission for less than 12 months prior to randomization. Subjects that had localized carcinoma (i.e., basal or squamous cell) of the skin which was resected for cure will not be excluded.
* FIP1 like 1-platelet derived growth factor receptor (FIP1L1-PDGFR) Status: Subjects who test positive for the FIP1L1-PDGFR fusion tyrosine kinase gene translocation.
* Subjects with chronic or ongoing active infections requiring systemic treatment, as well as subjects who have experienced clinically significant infections due to viruses, bacteria, and fungi within 4 weeks prior to randomization or subjects with a pre-existing helminthes infestation within 6 months prior to randomization
* Subjects with a known human immunodeficiency virus (e.g., HIV), other than that explained by the use of OCS or other therapy taken for HES.
* Other laboratory abnormalities: Evidence of clinically significant abnormality in the hematological, biochemical or urinalysis screen from the sample collected at screening, that could put the subject's safety at risk by participating in the study, as judged by the investigator
* Subjects who have previously received mepolizumab in the 4 months prior to randomization
* Subjects receiving intravenous or subcutaneous corticosteroids in the 4-week period prior to randomization or any other monoclonal antibodies within 30 days or 5 half-lives, whichever is longer, of randomization
* Subjects who have received treatment with an investigational agent (biologic or non-biologic) within the past 30 days or 5 drug half-lives whichever is longer, prior to randomization or subjects who are currently participating in any other interventional clinical study
* Subjects who are not responsive to oral corticosteroid based on clinical response or blood eosinophil counts
* Subjects with any history of hypersensitivity to any monoclonal antibody (including mepolizumab) or any steroid or steroid-containing product
* Subjects with a known or suspected history of alcohol or substance abuse at screening which in the opinion of the investigator could interfere with the subject's proper completion of the protocol requirement.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (41):
- United States (7):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Mayfield Heights, Ohio
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Salt Lake City, Utah
- Argentina (4):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Buenos Aires
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
- Brazil (4):
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Blumenau, Santa Catarina
  - GSK Investigational Site, Santo André - SP, São Paulo
  - GSK Investigational Site, Sorocaba, São Paulo
- France (4):
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Suresnes
  - GSK Investigational Site, Toulouse
- Germany (5):
  - GSK Investigational Site, Kirchheim -Teck, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
- Italy (2):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Florence, Tuscany
- Mexico (3):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Villahermosa, Tabasco
- Poland (2):
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
- Romania (3):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Târgu Mureş
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Roufosse F, Butterfield J, Steinfeld J, Bentley JH, von Maltzahn R, Kwon N, Nelsen L. Mepolizumab therapy improves the most bothersome symptoms in patients with hypereosinophilic syndrome. Front Med (Lausanne). 2023 Mar 29;10:1035250. doi: 10.3389/fmed.2023.1035250. eCollection 2023. PMID 37064032
- [Derived] Pane F, Lefevre G, Kwon N, Bentley JH, Yancey SW, Steinfeld J. Characterization of disease flares and impact of mepolizumab in patients with hypereosinophilic syndrome. Front Immunol. 2022 Aug 26;13:935996. doi: 10.3389/fimmu.2022.935996. eCollection 2022. PMID 36091012
- [Derived] Rothenberg ME, Roufosse F, Faguer S, Gleich GJ, Steinfeld J, Yancey SW, Mavropoulou E, Kwon N; HES Mepolizumab Study Group. Mepolizumab Reduces Hypereosinophilic Syndrome Flares Irrespective of Blood Eosinophil Count and Interleukin-5. J Allergy Clin Immunol Pract. 2022 Sep;10(9):2367-2374.e3. doi: 10.1016/j.jaip.2022.04.037. Epub 2022 May 12. PMID 35568330
- [Derived] Reiter A, Lefevre G, Cid MC, Kwon N, Mavropolou E, Yancey SW, Steinfeld J. Association Between Baseline Therapy and Flare Reduction in Mepolizumab-Treated Patients With Hypereosinophilic Syndrome. Front Immunol. 2022 Apr 13;13:840974. doi: 10.3389/fimmu.2022.840974. eCollection 2022. PMID 35493455
- [Derived] Gleich GJ, Roufosse F, Chupp G, Faguer S, Walz B, Reiter A, Yancey SW, Bentley JH, Steinfeld J; HES Mepolizumab Study Group. Safety and Efficacy of Mepolizumab in Hypereosinophilic Syndrome: An Open-Label Extension Study. J Allergy Clin Immunol Pract. 2021 Dec;9(12):4431-4440.e1. doi: 10.1016/j.jaip.2021.07.050. Epub 2021 Aug 10. PMID 34389506
- [Derived] Roufosse F, Kahn JE, Rothenberg ME, Wardlaw AJ, Klion AD, Kirby SY, Gilson MJ, Bentley JH, Bradford ES, Yancey SW, Steinfeld J, Gleich GJ; HES Mepolizumab study group. Efficacy and safety of mepolizumab in hypereosinophilic syndrome: A phase III, randomized, placebo-controlled trial. J Allergy Clin Immunol. 2020 Dec;146(6):1397-1405. doi: 10.1016/j.jaci.2020.08.037. Epub 2020 Sep 18. PMID 32956756

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This 32-week, randomized, double-blind, placebo-controlled study assessed the efficacy and safety of mepolizumab 300 milligrams (mg) subcutaneous (SC) every 4 weeks compared with placebo in adolescent and adult participants with severe hypereosinophilic syndrome (HES) receiving standard of care (SoC) therapy.
Pre-assignment Details: A total of 108 participants were enrolled in the study and randomized. The study was conducted in 13 countries.
Groups:
- Placebo: Participants were randomized to receive matching placebo SC every 4 weeks during the 32-Week treatment period while continuing their HES therapy. The final dose was administered at Week 28 with the completion of study treatment period achieved in the next 4-weekly visit.
- Mepolizumab 300 mg SC: Participants were randomized to receive 300 mg mepolizumab SC every 4 weeks during the 32-Week treatment period while continuing their HES therapy. The final dose was administered at Week 28 with the completion of study treatment period achieved in the next 4-weekly visit.
Period: Overall Study
Arm/Group | Placebo | Mepolizumab 300 mg SC
Started | 54 | 54
Completed | 52 | 52
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mepolizumab 300 mg SC | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.4 (18.25) | 46.6 (12.99) | 46.0 (15.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 30 | 57
  Male | 27 | 24 | 51
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian-Central/South Asian Heritage | 0 | 1 | 1
  Asian-East Asian Heritage | 1 | 0 | 1
  Asian-South East Asian Heritage | 1 | 0 | 1
  Black or African American | 2 | 0 | 2
  White-Arabic/North African Heritage | 1 | 0 | 1
  White-White/Caucasian/European Heritage | 47 | 52 | 99

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced an HES Flare or Who Withdrew From the Study During the 32-Week Study Treatment Period
Description: Percentage of participants who experienced >=1 HES flare during the 32-Week treatment period or who withdrew from the study has been presented. A HES flare is defined as a HES related clinical manifestation based on a physician-documented change in clinical signs or symptoms which resulted in need for an increase in the maintenance Oral Corticosteroid (OCS) dose by at least 10 mg per day for 5 days or an increase in or addition of any cytotoxic or immunosuppressive HES therapy. HES flare is also defined as receipt of two or more courses of blinded active OCS during the treatment period. Intent-to-treat (ITT) Population comprises of all randomized participants. This population was based on the treatment to which the participants were randomized. Any participant who received a treatment randomization number were considered to be randomized.
Time Frame: Up to Week 32
Population: ITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Mepolizumab 300 mg SC
Number analyzed (Participants) | 54 | 54
Percentage of participants | 56 | 28
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test stratified by Baseline oral corticosteroid (OCS) (0-<=20 mg per day and >20mg perday prednisone or equivalent) and region
Statistical Analysis 2: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.003, Regression, Logistic; Logistic regression analysis adjusted for Baseline OCS dose and region; Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.12 to 0.64] — Treatment comparison between placebo and mepolizumab 300 mg using odds ratio and 95% confidence interval (CI) has been presented. Odds ratio <1 indicated lower odds of HES flare with Mepolizumab compared with placebo

2. Secondary Outcome: Percentage of Participants Who Experienced a HES Flare or Who Withdrew From the Study During Week 20 Through Week 32
Description: HES flare during Week 20 through Week 32 was defined as a HES flare starting or ongoing on or after the date of the Week 20 visit up to and including the date of the Week 32 visit. Percentage of participants who experienced >=1 HES flare during Week 20 through Week 32 or who withdrew from the study has been presented.
Time Frame: Week 20 to Week 32
Population: ITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Mepolizumab 300 mg SC
Number analyzed (Participants) | 54 | 54
Percentage of participants | 35 | 17
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.020, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline OCS (0-<=20 mg per day and >20mg perday prednisone or equivalent) and region
Statistical Analysis 2: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.022, Regression, Logistic; Logistic regression analysis adjusted for Baseline OCS dose and region; Odds Ratio (OR) = 0.33, 95% CI 2-sided [0.13 to 0.85] — Treatment comparison between placebo and mepolizumab 300 mg using odds ratio and 95% CI has been presented. Odds ratio <1 indicated lower odds of HES flare with Mepolizumab compared with placebo

3. Secondary Outcome: Time to First HES Flare
Description: The time to first HES flare was calculated as (onset date of first HES flare minus date of first dose of study treatment) plus 1. Probability of first flare (by week 4, 8, 12, 16, 20, 24, 28, and 32) and corresponding 95% CI have been presented, calculated using the Kaplan-Meier method.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28 and 32
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: Probability expressed as percentage
Arm/Group | Placebo | Mepolizumab 300 mg SC
Number analyzed (Participants) | 54 | 54
Probability expressed as percentage
  Flares by Week 4 | 7.4 [2.8 to 18.5] | 5.6 [1.8 to 16.2]
  Flares by Week 8 | 14.9 [7.7 to 27.5] | 7.4 [2.8 to 18.5]
  Flares by Week 12 | 26.2 [16.4 to 40.2] | 9.3 [4.0 to 20.8]
  Flares by Week 16 | 33.8 [22.8 to 48.1] | 13.0 [6.4 to 25.3]
  Flares by Week 20 | 41.3 [29.5 to 55.7] | 13.0 [6.4 to 25.3]
  Flares by Week 24 | 48.9 [36.5 to 63.0] | 14.8 [7.7 to 27.4]
  Flares by Week 28 | 50.8 [38.3 to 64.8] | 20.5 [11.9 to 34.0]
  Flares by Week 32 | 52.7 [40.1 to 66.5] | 26.3 [16.5 to 40.3]
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.002, Regression, Cox — Cox proportional hazards regression analysis adjusted for Baseline OCS dose and region; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.18 to 0.67] — Treatment comparison between placebo and mepolizumab 300 mg using hazards ratio and its corresponding 95% CI has been presented. Hazard ratio <1 indicated a lower risk of HES flare with Mepolizumab compared with Placebo

4. Secondary Outcome: Number of HES Flares Per Participant Per Year
Description: The rate of HES flares for each participant was calculated as the number of observed HES flares divided by the time (expressed in years) between randomization and either the week 32 visit date if available, or the study withdrawal date. Negative binomial generalized linear model including Baseline OCS dose, region, treatment and observed time (offset variable). Wilcoxon test stratified by Baseline OCS (0-<=20mg/day, >20mg/day prednisone or equivalent) and region. Adjusted mean and 95% CI rate/year has been presented.
Time Frame: Up to Week 32
Population: ITT Population.
Measure: Mean (95% Confidence Interval); unit: Flares per participant per year
Arm/Group | Placebo | Mepolizumab 300 mg SC
Number analyzed (Participants) | 54 | 54
Flares per participant per year | 1.46 [1.05 to 2.02] | 0.50 [0.30 to 0.84]
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.002, Wilcoxon Rank Sum Test; Wilcoxon test stratified by Baseline OCS (0-<=20 mg/day, >20 mg/day prednisone or equivalent) and region; Rate Ratio = 0.34, 95% CI 2-sided [0.19 to 0.63] — Treatment comparison between placebo and mepolizumab 300 mg using rate ratio and 95% CI has been presented. Rate ratio <1 indicates a lower flare rate with Mepolizumab compared with Placebo

5. Secondary Outcome: Number of Participants With Change From Baseline in Fatigue Severity Based on Brief Fatigue Inventory (BFI) in Item 3 (Worst Level of Fatigue During Past 24 Hours) at Week 32 by Category
Description: The change from Baseline in fatigue severity (worst level of fatigue during past 24 hours) at Week 32 was calculated using the mean of the 7 daily assessments of BFI item 3 up to and including the date of the Week 32 visit as the Week 32 assessment, and the mean of the 7 daily assessments of BFI item 3 up to but not including the date of first dose of study treatment as the Baseline assessment. Wilcoxon Rank Sum test stratified by Baseline fatigue severity ("severe" defined as BFI item 3>=7 and "not severe" defined as BFI item 3<7), Baseline OCS (0-<=20mg/day and >20mg/day prednisone or equivalent) and region. Participants with missing change from Baseline at Week 32 were included in the worst category (>=4 point increase).
Time Frame: Baseline (Week 0) and at Week 32
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Mepolizumab 300 mg SC
Number analyzed (Participants) | 54 | 54
Participants
  >=4 point increase (>=3.5) | 7 | 5
  3 point increase (>=2.5 to <3.5) | 4 | 0
  2 point increase (>=1.5 to <2.5) | 4 | 5
  1 point increase (>=0.5 to <1.5) | 9 | 6
  No change (>-0.5 to <0.5) | 14 | 9
  1 point reduction (>-1.5 to <=-0.5) | 5 | 11
  2 point reduction (>-2.5 to <=-1.5) | 3 | 7
  3 point reduction (>-3.5 to <=-2.5) | 5 | 2
  >=4 point reduction (<=-3.5) | 3 | 9
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.036, Wilcoxon Rank Sum Test; P-value was calculated using Wilcoxon Rank Sum Test

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (non-SAEs) from start of study treatment until 28 days after last dose (Up to 32 weeks) are reported. Serious adverse events (SAEs) were collected from the day of randomization (Week 0) up to end of study (Up to Week 40).
Description: Non-SAEs and SAEs were collected for Safety Population. The Safety Population comprises of all participants who were randomized and who received at least one dose of study treatment.
Arm/Group | Placebo | Mepolizumab 300 mg SC
All-Cause Mortality (participants affected / at risk) | 0/54 | 1/54
Serious Adverse Events (participants affected / at risk) | 9/54 | 10/54
Other Adverse Events (participants affected / at risk) | 43/54 | 41/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=54) | Mepolizumab 300 mg SC (N=54)
Bronchitis (Infections and infestations) | 0 | 1
Bursitis infective (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=54) | Mepolizumab 300 mg SC (N=54)
Bronchitis (Infections and infestations) | 10 | 7
Nasopharyngitis (Infections and infestations) | 7 | 7
Rhinitis (Infections and infestations) | 6 | 5
Upper respiratory tract infection (Infections and infestations) | 2 | 8
Sinusitis (Infections and infestations) | 4 | 2
Urinary tract infection (Infections and infestations) | 0 | 5
Influenza (Infections and infestations) | 1 | 3
Oral herpes (Infections and infestations) | 2 | 2
Cystitis (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Arthritis infective (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 0
Onychomycosis (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 5
Vomiting (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 2
Toothache (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 5 | 3
Pyrexia (General disorders) | 2 | 4
Asthenia (General disorders) | 5 | 0
Influenza like illness (General disorders) | 2 | 3
Injection site reaction (General disorders) | 2 | 3
Peripheral swelling (General disorders) | 2 | 1
Malaise (General disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 7 | 7
Dizziness (Nervous system disorders) | 3 | 4
Hypoaesthesia (Nervous system disorders) | 1 | 3
Paraesthesia (Nervous system disorders) | 0 | 3
Presyncope (Nervous system disorders) | 3 | 0
Somnolence (Nervous system disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Hypertension (Vascular disorders) | 2 | 1
Palpitations (Cardiac disorders) | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-04-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT02836496/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT02836496/SAP_001.pdf